CLINICAL TRIAL: NCT05628025
Title: Simulation-Based Enucleation Training: Initial Experience Using 3D-printed Organ Phantoms
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-10107
Record Dates: First submitted 2021-09-13; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: BPH
Keywords: Simulator; Training; Laser Enucleation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trainees: Residents in urology or urologists with little LEP experience. Trainee group will be stratified by level of experience.
  Interventions: Other: Organ phantom of prostate
- Experts: Urologists with at least 5 years LEP experience.
  Interventions: Other: Organ phantom of prostate

INTERVENTIONS:
Other: Organ phantom of prostate — Participants will operate on a 3D printed model of the prostate.

SUMMARY:
There are many possible surgical treatments when a patient presents with lower urinary tract symptoms due to an enlarged prostate, termed benign prostatic hyperplasia or BPH. One technique consists of using a laser to remove prostatic tissue through the penis, called laser enucleation of the prostate or LEP. LEP also has excellent properties to reduce blood loss and results in shorter hospital stays. Trainees must observe and perform several procedures before mastering the LEP technique. Different models have been used to mimic the LEP experience for surgeon trainees, such as virtual simulators or synthetic models. While these simulators offer an alternative to LEP procedures on real patients, they may lack realism which renders the simulator less representative than the real procedure.The 3D-printed prostate model of the present study mimics the properties of real-life prostatic tissue. In the setting of the MasterClass, trainees will perform LEP on the 3D models under the supervision of three experts. While the 3D organ phantom has been used to practice performing other procedures, this is the first time it will evaluated for LEP training. For this reason, the investigators will be assessing this model as a training tool.

DETAILED DESCRIPTION:
Numerous surgical treatment options exist for benign prostatic hyperplasia (BPH). Laser enucleation of the prostate (LEP) was introduced in the therapeutic arsenal about twenty years ago, and has become a popular treatment due to its excellent hemostatic properties. Moreover, LEP is associated with less blood loss and shorter hospital stays. One disadvantage however may be the longer learning curve for trainees compared to transurethral resection of the prostate (TURP), which is the current gold standard for treatment.

It is estimated that a surgeon can safely and efficiently perform holmium LEP after about 50 cases. Simulator-based training has been widely proposed as a training tool for surgeons to learn LEP. Integrating simulators in surgical training allows surgeons to develop skills in LEP without negative consequences on real patients. Simulators range from virtual reality to synthetic bench models, and all face the same challenge of creating a realistic experience that accurately mimics real-life LEP, and helps surgeons develop skills they can transfer to the operating room.

The prostate organ phantom in the present study is composed of hydrogels and uses 3D molds to recreate prostatic tissue and anatomy. This model has successfully been used to practice TURP procedures, however has not yet been validated for LEP training. This observational, prospective and comparative study aims to validate the 3D prostate organ for LEP training. In the setting of a MasterClass, trainees will perform LEP on two 3D models under the supervision of three experts in LEP. The content and face validity of the organ phantoms will be evaluated by the MasterClass participants through a questionnaire. Performance outcomes of trainees will also be collected by visually examining the models and weighing the models pre- and post-operatively. By validating this simulator for LEP training, the investigators hope to elucidate the role of simulators, and specifically the role of a 3D organ phantom, in future training programs.

ELIGIBILITY:
Inclusion Criteria:

* Participate in LEP MasterClass

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Urologists in training seeking to improve skills in LEP and experts in LEP.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Content and face validity of the organ phantom model in LEP training. | Up to one year post-workshop
  Assessed with validated questionnaire using a Likert scale.

SECONDARY OUTCOMES:
Verify the reproducibility of each 3D printed model. | Up to one year post-workshop
  Assessed with validated questionnaire using a Likert scale.
Determine the surgical performance outcomes of trainees based on level of expertise, and compared with LEP experts (construct validity). | Up to one year post-workshop
  Percentage of prostatic tissue resected.
Assess the perceived difficulty of each step of LEP by trainees. | Up to one year post-workshop
  Assessed with validated questionnaire using a Likert scale.
Gauge the feasibility and acceptability of integrating simulators in LEP training. | Up to one year post-workshop
  Assessed with validated questionnaire using a Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Canada

IPD SHARING:
Plan to Share IPD: Undecided